CLINICAL TRIAL: NCT03364036
Title: A 2-year Prospective Study to Evaluate the Onset of Action of Mavenclad® in Subjects With Highly Active Relapsing Multiple Sclerosis (MAGNIFY)
Brief Title: Evaluation of the Onset of Action in Highly Active MS (MAGNIFY)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS700568_0022; 2017-002631-42 (EudraCT Number)
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Mavenclad ®; Cladribine
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mavenclad® (Experimental)
  Interventions: Drug: Mavenclad®

INTERVENTIONS:
Drug: Mavenclad® — Participants received Mavenclad® 3.5 milligram per kilogram (mg/kg) of body weight over 2 years, administered as 1 treatment course of 1.75 mg/kg per year.
  Other Names: Cladribine

SUMMARY:
The main purpose of the study was to determine the onset of Mavenclad® action by frequent magnetic resonance imaging (MRI) assessment of the combined unique active (CUA) lesions in participants with highly active relapsing multiple sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Highly active RMS as defined by:
* One relapse in the previous year and at least 1 T1 Gadolinium (Gd)+ lesion or 9 or more T2 lesions, while on therapy with other disease modifying drugs (DMDs)
* Two or more relapses in the previous year, whether on DMD treatment or not.
* Expanded Disability Status Scale (EDSS) score less than equals to (<=) 5.0.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Previous exposure to drugs such as fingolimod, natalizumab, alemtuzumab, mitoxantrone and ocrelizumab.
* Positive hepatitis C or hepatitis B surface antigen test and/or hepatits B core antibody test for immunoglobulin G (IgG) and/or immunoglobulin M (IgM).
* Current or previous history of immune deficiency disorders including a positive human immunodeficiency virus (HIV) result.
* Currently receiving immunosuppressive or myelosuppressive therapy with, for example, monoclonal antibodies, methotrexate, cyclophosphamide, cyclosporine or azathioprine, or chronic use of corticosteroids.
* History of tuberculosis , presence of active tuberculosis, or latent tuberculosis
* Evidence or suspect of Progressive Multifocal Leukoencephalopathy (PML) in Magnetic Resonance Imaging (MRI).
* Active malignancy or history of malignancy.
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (54):
- Australia (4):
  - Liverpool Hospital, Sydney, New South Wales
  - John Hunter Hospital, Hunter Region Mail Centre
  - Perron Institute - Neurology, Nedlands
  - The Alfred Hospital, Prahran
- Austria (2):
  - Klagenfurt1, Klagenfurt
  - Paracelsus Medical University Salzburg, Salzburg
- Canada (4):
  - MS Clinical Trials Group, Vancouver, British Columbia
  - UB - State University of New York, London, Ontario
  - University of Alberta, Edmonton
  - Montreal Neurological Hospital, Montreal
- Czechia (5):
  - Fakultni nemocnice Brno, Brno-Bohunice, Brno-Bohunice
  - Nemocnice Pardubickeho kraje, a.s. Pardubicka nemocnice, Pardubice, Pardubický kraj
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - FN Hradec Kralove, Choceň
  - Fakultni nemocnice v Motole, Prague
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - FinnMedi Oy vastaanotto - Finn-Medi 3, Tampere
  - Turku University Hospital, Turku
- France (7):
  - CHU de Pontchaillou, Rennes, Ille Et Vilaine
  - CHRU de Lille, Lille
  - CHU Nice - Hôpital Pasteur, Nice
  - CHU Montpellier-Nîmes - Hôpital Caremeau, Nîmes
  - CHU Nîmes, Nîmes
  - CHU de Poissy, Poissy
  - Hôpital Civil, Strasbourg
- Germany (8):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Neuro Centrum Science GmbH, Erbach im Odenwald
  - Universitätsklinikum Essen, Essen
  - Neurologische Praxis Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
- Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpo, Szeged, Hungary
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Rambam MC, Haifa
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - Policlinico Universitario SS Annunziata, Chieti
  - Seconda Univesità degli Studi di Napoli, AOU, Napoli
  - IRCSS Neuromed Istituto Neurologico Mediterraneo, Roma
  - Universita di SIENA, Siena
- Poland (3):
  - Indywidualna Praktyka Lekarska Prof. Konrad Rejdak, Lublin, Lublin Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 7 SUM, Katowice
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Stanislawa Szyszko SUM w Katowicach, Zabrze
- Spain (5):
  - Hospital de Cruces, Baracaldo Vizcaya, Vizcaya
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Vithas NISA Sevilla, Seville
  - Hospital La Fe, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhus, Gothenburg
  - Akademiskt Specialist Centrum - Centrum för Neurologi, plan 5, Stockholm
- United Kingdom (3):
  - University Hospital of Wales, Cardiff, Wales
  - Queen Elizabeth Hospital, Birmingham
  - Sheffield Teaching Hospitals Sheffield, Sheffield

REFERENCES:
- [Result] de Stefano N, Barkhof F, Montalban X, Achiron A, Derfuss T, Chan A, Hodgkinson S, Prat A, Leocani L, Schmierer K, Sellebjerg F, Vermersch P, Wiendl H, Keller B, Roy S; MAGNIFY-MS Study Group. Early Reduction of MRI Activity During 6 Months of Treatment With Cladribine Tablets for Highly Active Relapsing Multiple Sclerosis: MAGNIFY-MS. Neurol Neuroimmunol Neuroinflamm. 2022 Jun 14;9(4):e1187. doi: 10.1212/NXI.0000000000001187. Print 2022 Jul. PMID 35701185
- [Derived] Schmierer K, Wiendl H, Barkhof F, Montalban X, Achiron A, Derfuss T, Chan A, Hodgkinson S, Prat A, Leocani L, Sellebjerg F, Vermersch P, Jin H, Sponton L, Chudecka A, Gardner L, De Stefano N. Clinical and mechanistic effects of cladribine in relapsing multiple sclerosis: 2-year results from the MAGNIFY-MS Study. Ther Adv Neurol Disord. 2025 Jul 31;18:17562864251351760. doi: 10.1177/17562864251351760. eCollection 2025. PMID 40756532
- [Derived] Wiendl H, Barkhof F, Montalban X, Achiron A, Derfuss T, Chan A, Hodgkinson S, Prat A, Leocani L, Schmierer K, Sellebjerg F, Vermersch P, Jin H, Chudecka A, Kloetgen A, Lin D, Gardner L, De Stefano N. Blood biomarker dynamics in people with relapsing multiple sclerosis treated with cladribine tablets: results of the 2-year MAGNIFY-MS study. Front Immunol. 2025 Feb 3;16:1512189. doi: 10.3389/fimmu.2025.1512189. eCollection 2025. PMID 39963134
- [Derived] Wiendl H, Schmierer K, Hodgkinson S, Derfuss T, Chan A, Sellebjerg F, Achiron A, Montalban X, Prat A, De Stefano N, Barkhof F, Leocani L, Vermersch P, Chudecka A, Mwape C, Holmberg KH, Boschert U, Roy S; MAGNIFY-MS Study Group. Specific Patterns of Immune Cell Dynamics May Explain the Early Onset and Prolonged Efficacy of Cladribine Tablets: A MAGNIFY-MS Substudy. Neurol Neuroimmunol Neuroinflamm. 2022 Nov 21;10(1):e200048. doi: 10.1212/NXI.0000000000200048. Print 2023 Jan. PMID 36411081
- [Derived] Schmierer K, Wiendl H, Oreja-Guevara C, Centonze D, Chudecka A, Roy S, Boschert U. Varicella zoster virus and influenza vaccine antibody titres in patients from MAGNIFY-MS who were treated with cladribine tablets for highly active relapsing multiple sclerosis. Mult Scler. 2022 Nov;28(13):2151-2153. doi: 10.1177/13524585221099413. Epub 2022 Jun 7. No abstract available. PMID 35672923
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0022
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 270 participants were enrolled in the study from different trial sites across14 countries (Austria, Germany, Hungary, Poland, Czechia, Italy, Spain, France, United Kingdom of Great Britain and Northern Ireland, Finland, Sweden, Israel, Australia and Canada).
Groups:
- Experimental: Mavenclad®: Participants received Mavenclad® 3.5 milligram per kilogram (mg/kg) of body weight over 2 years, administered as 1 treatment course of 1.75 mg/kg per year.
Period: Overall Study
Arm/Group | Experimental: Mavenclad®
Started | 270
Full Analysis Set (FAS) | 270
Completed | 270
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants from the intent-to-treat (ITT [ITT population included all participants classified as eligible]) set who received at least one dose of the study treatment.
Arm/Group | Experimental: Mavenclad®
Number analyzed (Participants) | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 246
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Other: American Indian or Alaska Native | 0
  Other: Asian | 2
  Other: Native Hawaiian or Other Pacific Islander | 0
  Other: Black or African American | 1
  Other: White | 225
  Other: More than one race | 12
  Other: Unknown or Not Reported | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Period (Period Screening to Baseline) in Counts of Combined Unique Active (CUA) Magnetic Resonance Imaging (MRI) Lesions at Period 1 (Month 1-6)
Description: CUA lesions were measured by using MRI scans.
Time Frame: Baseline period (the period screening to Baseline), Period 1 (Month 1-6)
Population: FAS included all participants from the ITT set who received at least one dose of the study treatment. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Experimental: Mavenclad®
Number analyzed (Participants) | 252
lesions | -1.211 (3.4413)

2. Primary Outcome: Change From Baseline Period (Period Screening to Baseline) in Counts of Combined Unique Active (CUA) Magnetic Resonance Imaging (MRI) Lesions at Period 2 (Month 2-6)
Description: CUA lesions were measured by using MRI scans.
Time Frame: Baseline period (the period screening to Baseline), Period 2 (Month 2-6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Experimental: Mavenclad®
Number analyzed (Participants) | 252
lesions | -1.521 (4.0558)

3. Primary Outcome: Change From Baseline Period (Period Screening to Baseline) in Counts of Combined Unique Active (CUA) Magnetic Resonance Imaging (MRI) Lesions at Period 3 (Month 3-6)
Description: CUA lesions were measured by using MRI scans.
Time Frame: Baseline period (the period screening to Baseline), Period 3 (Month 3-6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Experimental: Mavenclad®
Number analyzed (Participants) | 246
lesions | -1.499 (3.4244)

4. Secondary Outcome: Percent Change From Baseline in Counts of Immune Cell Subsets - B Cells at Month 3, 6, 12, 15, 18 and 24
Description: B cell population counts are: CD19 B cells (TBNK panel), CD20 B cells (B cell panel), Memory B cells (B cell panel), Activated B cells (B cell panel), Total plasma cells (B cell panel), Short-lived plasma cells (B cell panel), Naïve B cells (B cell panel), Transitional B cells (B cell panel), and Regulatory B cells (B cell panel).
Time Frame: Baseline, Month 3, 6, 12, 15, 18 and 24
Population: FAS included all participants from the ITT set who received at least one dose of the study treatment. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specified categories.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Experimental: Mavenclad®
Number analyzed (Participants) | 204
Percent change
  CD19 B cells (TBNK panel), Month 3 | -80.14 [-85.85 to -73.65]
  CD19 B cells (TBNK panel), Month 6: number analyzed (Participants) | 200
  CD19 B cells (TBNK panel), Month 6 | -60.60 [-72.43 to -45.62]
  CD19 B cells (TBNK panel), Month 12: number analyzed (Participants) | 195
  CD19 B cells (TBNK panel), Month 12 | -26.88 [-46.67 to -3.70]
  CD19 B cells (TBNK panel), Month 15: number analyzed (Participants) | 161
  CD19 B cells (TBNK panel), Month 15 | -77.24 [-85.64 to -65.59]
  CD19 B cells (TBNK panel), Month 18: number analyzed (Participants) | 163
  CD19 B cells (TBNK panel), Month 18 | -55.30 [-69.55 to -39.30]
  CD19 B cells (TBNK panel), Month 24: number analyzed (Participants) | 172
  CD19 B cells (TBNK panel), Month 24 | -27.65 [-46.11 to 1.77]
  CD20 B cells (B cell panel), Month 3: number analyzed (Participants) | 200
  CD20 B cells (B cell panel), Month 3 | -80.50 [-86.46 to -74.23]
  CD20 B cells (B cell panel), Month 6: number analyzed (Participants) | 196
  CD20 B cells (B cell panel), Month 6 | -60.32 [-71.94 to -43.77]
  CD20 B cells (B cell panel), Month 12: number analyzed (Participants) | 191
  CD20 B cells (B cell panel), Month 12 | -24.56 [-45.77 to -2.54]
  CD20 B cells (B cell panel), Month 15: number analyzed (Participants) | 159
  CD20 B cells (B cell panel), Month 15 | -77.11 [-85.54 to -65.25]
  CD20 B cells (B cell panel), Month 18: number analyzed (Participants) | 163
  CD20 B cells (B cell panel), Month 18 | -54.21 [-68.62 to -36.91]
  CD20 B cells (B cell panel), Month 24: number analyzed (Participants) | 169
  CD20 B cells (B cell panel), Month 24 | -24.77 [-43.43 to 8.84]
  Memory B cells (B cell panel), Month 3: number analyzed (Participants) | 200
  Memory B cells (B cell panel), Month 3 | -92.69 [-95.56 to -88.52]
  Memory B cells (B cell panel), Month 6: number analyzed (Participants) | 196
  Memory B cells (B cell panel), Month 6 | -91.56 [-94.14 to -86.80]
  Memory B cells (B cell panel), Month 12: number analyzed (Participants) | 189
  Memory B cells (B cell panel), Month 12 | -86.90 [-91.57 to -80.14]
  Memory B cells (B cell panel), Month 15: number analyzed (Participants) | 159
  Memory B cells (B cell panel), Month 15 | -96.47 [-97.75 to -93.25]
  Memory B cells (B cell panel), Month 18: number analyzed (Participants) | 162
  Memory B cells (B cell panel), Month 18 | -94.67 [-96.70 to -91.41]
  Memory B cells (B cell panel), Month 24: number analyzed (Participants) | 169
  Memory B cells (B cell panel), Month 24 | -89.29 [-93.61 to -84.91]
  Activated B cells (B cell panel), Month 3: number analyzed (Participants) | 200
  Activated B cells (B cell panel), Month 3 | -74.02 [-83.29 to -61.45]
  Activated B cells (B cell panel), Month 6: number analyzed (Participants) | 196
  Activated B cells (B cell panel), Month 6 | -60.91 [-74.77 to -38.25]
  Activated B cells (B cell panel), Month 12: number analyzed (Participants) | 190
  Activated B cells (B cell panel), Month 12 | -28.82 [-52.68 to -1.85]
  Activated B cells (B cell panel), Month 15: number analyzed (Participants) | 159
  Activated B cells (B cell panel), Month 15 | -73.02 [-83.81 to -62.22]
  Activated B cells (B cell panel), Month 18: number analyzed (Participants) | 163
  Activated B cells (B cell panel), Month 18 | -51.87 [-65.00 to -28.54]
  Activated B cells (B cell panel), Month 24: number analyzed (Participants) | 169
  Activated B cells (B cell panel), Month 24 | -15.95 [-40.82 to 29.33]
  Total plasma cells (B cell panel), Month 3: number analyzed (Participants) | 200
  Total plasma cells (B cell panel), Month 3 | -66.62 [-82.38 to -33.69]
  Total plasma cells (B cell panel), Month 6: number analyzed (Participants) | 196
  Total plasma cells (B cell panel), Month 6 | -59.00 [-78.63 to -28.51]
  Total plasma cells (B cell panel), Month 12: number analyzed (Participants) | 190
  Total plasma cells (B cell panel), Month 12 | -54.75 [-71.43 to -19.03]
  Total plasma cells (B cell panel), Month 15: number analyzed (Participants) | 155
  Total plasma cells (B cell panel), Month 15 | -78.02 [-89.68 to -60.13]
  Total plasma cells (B cell panel), Month 18: number analyzed (Participants) | 158
  Total plasma cells (B cell panel), Month 18 | -72.39 [-84.71 to -57.31]
  Total plasma cells (B cell panel), Month 24: number analyzed (Participants) | 167
  Total plasma cells (B cell panel), Month 24 | -62.47 [-80.79 to -36.26]
  Short-lived plasma cells (B cell panel), Month 3: number analyzed (Participants) | 200
  Short-lived plasma cells (B cell panel), Month 3 | -68.18 [-84.72 to -43.46]
  Short-lived plasma cells (B cell panel), Month 6: number analyzed (Participants) | 195
  Short-lived plasma cells (B cell panel), Month 6 | -56.55 [-77.83 to -31.98]
  Short-lived plasma cells (B cell panel), Month 12: number analyzed (Participants) | 188
  Short-lived plasma cells (B cell panel), Month 12 | -56.70 [-76.20 to -23.22]
  Short-lived plasma cells (B cell panel), Month 15: number analyzed (Participants) | 158
  Short-lived plasma cells (B cell panel), Month 15 | -82.96 [-93.23 to -69.90]
  Short-lived plasma cells (B cell panel), Month 18: number analyzed (Participants) | 161
  Short-lived plasma cells (B cell panel), Month 18 | -79.54 [-90.76 to -65.70]
  Short-lived plasma cells (B cell panel), Month 24: number analyzed (Participants) | 168
  Short-lived plasma cells (B cell panel), Month 24 | -70.10 [-83.17 to -45.12]
  Naïve B cells (B cell panel), Month 3: number analyzed (Participants) | 200
  Naïve B cells (B cell panel), Month 3 | -75.87 [-84.21 to -66.18]
  Naïve B cells (B cell panel), Month 6: number analyzed (Participants) | 196
  Naïve B cells (B cell panel), Month 6 | -45.87 [-61.72 to -24.82]
  Naïve B cells (B cell panel), Month 12: number analyzed (Participants) | 189
  Naïve B cells (B cell panel), Month 12 | 1.63 [-20.85 to 35.59]
  Naïve B cells (B cell panel), Month 15: number analyzed (Participants) | 159
  Naïve B cells (B cell panel), Month 15 | -69.17 [-79.40 to -51.59]
  Naïve B cells (B cell panel), Month 18: number analyzed (Participants) | 162
  Naïve B cells (B cell panel), Month 18 | -39.73 [-57.61 to -5.27]
  Naïve B cells (B cell panel), Month 24: number analyzed (Participants) | 169
  Naïve B cells (B cell panel), Month 24 | 10.85 [-21.00 to 45.19]
  Transitional B cells (B cell panel), Month 3: number analyzed (Participants) | 200
  Transitional B cells (B cell panel), Month 3 | -4.06 [-38.65 to 56.25]
  Transitional B cells (B cell panel), Month 6: number analyzed (Participants) | 196
  Transitional B cells (B cell panel), Month 6 | 14.82 [-28.68 to 63.34]
  Transitional B cells (B cell panel), Month 12: number analyzed (Participants) | 191
  Transitional B cells (B cell panel), Month 12 | 11.92 [-26.75 to 64.99]
  Transitional B cells (B cell panel), Month 15: number analyzed (Participants) | 159
  Transitional B cells (B cell panel), Month 15 | 28.69 [-29.88 to 92.02]
  Transitional B cells (B cell panel), Month 18: number analyzed (Participants) | 163
  Transitional B cells (B cell panel), Month 18 | 11.27 [-22.94 to 67.22]
  Transitional B cells (B cell panel), Month 24: number analyzed (Participants) | 170
  Transitional B cells (B cell panel), Month 24 | 6.30 [-27.06 to 69.12]
  Regulatory B cells (B cell panel), Month 3: number analyzed (Participants) | 200
  Regulatory B cells (B cell panel), Month 3 | 110.73 [17.78 to 290.50]
  Regulatory B cells (B cell panel), Month 6: number analyzed (Participants) | 196
  Regulatory B cells (B cell panel), Month 6 | 92.95 [19.07 to 231.41]
  Regulatory B cells (B cell panel), Month 12: number analyzed (Participants) | 191
  Regulatory B cells (B cell panel), Month 12 | 30.64 [-18.33 to 134.17]
  Regulatory B cells (B cell panel), Month 15: number analyzed (Participants) | 159
  Regulatory B cells (B cell panel), Month 15 | 91.57 [15.05 to 288.71]
  Regulatory B cells (B cell panel), Month 18: number analyzed (Participants) | 163
  Regulatory B cells (B cell panel), Month 18 | 33.83 [-21.55 to 150.29]
  Regulatory B cells (B cell panel), Month 24: number analyzed (Participants) | 170
  Regulatory B cells (B cell panel), Month 24 | 1.62 [-36.85 to 98.81]

5. Secondary Outcome: Percent Change From Baseline in Counts of Immune Cell Subsets - T Cells at Month 3, 6, 12, 15, 18 and 24
Description: T cell population counts are: Total CD4 T cells (TBNK panel), CD4 Th1 cells (T cell panel), CD4 Th17 T cells (T cell panel), CD4 Regulatory T cells (T cell panel), and Total CD8 T cells (TBNK panel).
Time Frame: Baseline, Month 3, 6, 12, 15, 18 and 24
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Experimental: Mavenclad®
Number analyzed (Participants) | 204
Percent change
  Total CD4 T cells (TBNK panel), Month 3 | -48.60 [-62.55 to -37.05]
  Total CD4 T cells (TBNK panel), Month 6: number analyzed (Participants) | 200
  Total CD4 T cells (TBNK panel), Month 6 | -47.18 [-59.72 to -34.68]
  Total CD4 T cells (TBNK panel), Month 12: number analyzed (Participants) | 195
  Total CD4 T cells (TBNK panel), Month 12 | -40.16 [-55.59 to -27.74]
  Total CD4 T cells (TBNK panel), Month 15: number analyzed (Participants) | 161
  Total CD4 T cells (TBNK panel), Month 15 | -69.04 [-79.78 to -58.61]
  Total CD4 T cells (TBNK panel), Month 18: number analyzed (Participants) | 163
  Total CD4 T cells (TBNK panel), Month 18 | -66.98 [-75.03 to -55.24]
  Total CD4 T cells (TBNK panel), Month 24: number analyzed (Participants) | 172
  Total CD4 T cells (TBNK panel), Month 24 | -57.51 [-67.54 to -47.47]
  CD4 Th1 cells (T cell panel), Month 3: number analyzed (Participants) | 203
  CD4 Th1 cells (T cell panel), Month 3 | -44.35 [-61.62 to -30.01]
  CD4 Th1 cells (T cell panel), Month 6: number analyzed (Participants) | 197
  CD4 Th1 cells (T cell panel), Month 6 | -43.20 [-56.95 to -28.94]
  CD4 Th1 cells (T cell panel), Month 12: number analyzed (Participants) | 192
  CD4 Th1 cells (T cell panel), Month 12 | -35.55 [-50.76 to -17.71]
  CD4 Th1 cells (T cell panel), Month 15: number analyzed (Participants) | 159
  CD4 Th1 cells (T cell panel), Month 15 | -63.68 [-77.41 to -51.43]
  CD4 Th1 cells (T cell panel), Month 18: number analyzed (Participants) | 163
  CD4 Th1 cells (T cell panel), Month 18 | -63.01 [-74.41 to -49.62]
  CD4 Th1 cells (T cell panel), Month 24: number analyzed (Participants) | 170
  CD4 Th1 cells (T cell panel), Month 24 | -52.86 [-62.71 to -40.22]
  CD4 Th17 T cells (T cell panel), Month 3: number analyzed (Participants) | 200
  CD4 Th17 T cells (T cell panel), Month 3 | -33.09 [-53.72 to -15.56]
  CD4 Th17 T cells (T cell panel), Month 6: number analyzed (Participants) | 193
  CD4 Th17 T cells (T cell panel), Month 6 | -30.26 [-46.84 to -10.70]
  CD4 Th17 T cells (T cell panel), Month 12: number analyzed (Participants) | 185
  CD4 Th17 T cells (T cell panel), Month 12 | -18.39 [-38.10 to 10.51]
  CD4 Th17 T cells (T cell panel), Month 15: number analyzed (Participants) | 152
  CD4 Th17 T cells (T cell panel), Month 15 | -44.57 [-59.51 to -28.43]
  CD4 Th17 T cells (T cell panel), Month 18: number analyzed (Participants) | 157
  CD4 Th17 T cells (T cell panel), Month 18 | -42.77 [-55.47 to -18.37]
  CD4 Th17 T cells (T cell panel), Month 24: number analyzed (Participants) | 164
  CD4 Th17 T cells (T cell panel), Month 24 | -31.74 [-46.81 to -3.84]
  CD4 Regulatory T cells (T cell panel), Month 3: number analyzed (Participants) | 203
  CD4 Regulatory T cells (T cell panel), Month 3 | -25.98 [-42.82 to -11.42]
  CD4 Regulatory T cells (T cell panel), Month 6: number analyzed (Participants) | 197
  CD4 Regulatory T cells (T cell panel), Month 6 | -29.84 [-41.82 to -11.66]
  CD4 Regulatory T cells (T cell panel), Month 12: number analyzed (Participants) | 192
  CD4 Regulatory T cells (T cell panel), Month 12 | -25.60 [-38.18 to -10.45]
  CD4 Regulatory T cells (T cell panel), Month 15: number analyzed (Participants) | 159
  CD4 Regulatory T cells (T cell panel), Month 15 | -48.40 [-59.80 to -35.82]
  CD4 Regulatory T cells (T cell panel), Month 18: number analyzed (Participants) | 163
  CD4 Regulatory T cells (T cell panel), Month 18 | -48.73 [-60.71 to -34.86]
  CD4 Regulatory T cells (T cell panel), Month 24: number analyzed (Participants) | 169
  CD4 Regulatory T cells (T cell panel), Month 24 | -40.30 [-52.78 to -27.15]
  Total CD8 T cells (TBNK panel), Month 3 | -42.33 [-54.55 to -22.17]
  Total CD8 T cells (TBNK panel), Month 6: number analyzed (Participants) | 200
  Total CD8 T cells (TBNK panel), Month 6 | -39.42 [-52.98 to -19.88]
  Total CD8 T cells (TBNK panel), Month 12: number analyzed (Participants) | 195
  Total CD8 T cells (TBNK panel), Month 12 | -36.28 [-51.42 to -15.79]
  Total CD8 T cells (TBNK panel), Month 15: number analyzed (Participants) | 161
  Total CD8 T cells (TBNK panel), Month 15 | -57.08 [-69.20 to -38.74]
  Total CD8 T cells (TBNK panel), Month 18: number analyzed (Participants) | 163
  Total CD8 T cells (TBNK panel), Month 18 | -54.44 [-67.77 to -35.12]
  Total CD8 T cells (TBNK panel), Month 24: number analyzed (Participants) | 172
  Total CD8 T cells (TBNK panel), Month 24 | -45.93 [-58.41 to -30.17]

6. Secondary Outcome: Percent Change From Baseline in Counts of Immune Cell Subsets - NK Cells at Month 3, 6, 12, 15, 18 and 24
Description: NK cell population counts are: CD16+ CD56+ NK Cells, CD16+ NK Cells, NK p46 cells, CD16lowCD56bright, and CD16brightCD56dim.
Time Frame: Baseline, Month 3, 6, 12, 15, 18 and 24.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Experimental: Mavenclad®
Number analyzed (Participants) | 203
Percent change
  CD16+ CD56- NK cells, Month 3 | 3.08 [-32.82 to 48.59]
  CD16+ CD56- NK cells, Month 6: number analyzed (Participants) | 197
  CD16+ CD56- NK cells, Month 6 | -8.88 [-35.60 to 40.41]
  CD16+ CD56- NK cells, Month 12: number analyzed (Participants) | 192
  CD16+ CD56- NK cells, Month 12 | 9.44 [-38.02 to 65.90]
  CD16+ CD56- NK cells, Month 15: number analyzed (Participants) | 159
  CD16+ CD56- NK cells, Month 15 | 27.70 [-24.44 to 104.4]
  CD16+ CD56- NK cells, Month 18: number analyzed (Participants) | 163
  CD16+ CD56- NK cells, Month 18 | 7.89 [-31.60 to 55.64]
  CD16+ CD56- NK cells, Month 24: number analyzed (Participants) | 170
  CD16+ CD56- NK cells, Month 24 | -21.64 [-50.92 to 38.15]
  CD16+ NK cells, Month 3 | -32.50 [-49.49 to -12.61]
  CD16+ NK cells, Month 6: number analyzed (Participants) | 197
  CD16+ NK cells, Month 6 | -21.78 [-44.93 to 1.81]
  CD16+ NK cells, Month 12: number analyzed (Participants) | 192
  CD16+ NK cells, Month 12 | -8.10 [-33.88 to 14.37]
  CD16+ NK cells, Month 15: number analyzed (Participants) | 159
  CD16+ NK cells, Month 15 | -28.56 [-48.73 to -4.90]
  CD16+ NK cells, Month 18: number analyzed (Participants) | 163
  CD16+ NK cells, Month 18 | -21.47 [-40.28 to 2.74]
  CD16+ NK cells, Month 24: number analyzed (Participants) | 170
  CD16+ NK cells, Month 24 | -13.76 [-35.92 to 12.58]
  NK p46 cells, Month 3 | -20.85 [-47.77 to 17.63]
  NK p46 cells, Month 6: number analyzed (Participants) | 197
  NK p46 cells, Month 6 | -22.38 [-45.67 to 21.71]
  NK p46 cells, Month 12: number analyzed (Participants) | 192
  NK p46 cells, Month 12 | 29.49 [-18.73 to 116.77]
  NK p46 cells, Month 15: number analyzed (Participants) | 158
  NK p46 cells, Month 15 | 28.42 [-11.69 to 97.64]
  NK p46 cells, Month 18: number analyzed (Participants) | 163
  NK p46 cells, Month 18 | 71.73 [2.68 to 154.75]
  NK p46 cells, Month 24: number analyzed (Participants) | 170
  NK p46 cells, Month 24 | 77.70 [18.42 to 175.01]
  CD16low CD56bright, Month 3 | -8.94 [-36.65 to 31.46]
  CD16low CD56bright, Month 6: number analyzed (Participants) | 197
  CD16low CD56bright, Month 6 | 3.72 [-26.06 to 42.24]
  CD16low CD56bright, Month 12: number analyzed (Participants) | 192
  CD16low CD56bright, Month 12 | 2.56 [-20.62 to 41.41]
  CD16low CD56bright, Month 15: number analyzed (Participants) | 159
  CD16low CD56bright, Month 15 | 4.77 [-23.35 to 49.22]
  CD16low CD56bright, Month 18: number analyzed (Participants) | 163
  CD16low CD56bright, Month 18 | 30.13 [-8.52 to 75.67]
  CD16low CD56bright, Month 24: number analyzed (Participants) | 170
  CD16low CD56bright, Month 24 | 17.21 [-20.09 to 82.09]
  CD16bright CD56dim, Month 3 | -36.13 [-55.16 to -14.13]
  CD16bright CD56dim, Month 6: number analyzed (Participants) | 197
  CD16bright CD56dim, Month 6 | -25.61 [-46.87 to 1.97]
  CD16bright CD56dim, Month 12: number analyzed (Participants) | 192
  CD16bright CD56dim, Month 12 | -11.05 [-38.53 to 16.63]
  CD16bright CD56dim, Month 15: number analyzed (Participants) | 159
  CD16bright CD56dim, Month 15 | -35.05 [-55.45 to -8.85]
  CD16bright CD56dim, Month 18: number analyzed (Participants) | 163
  CD16bright CD56dim, Month 18 | -24.99 [-45.87 to -0.29]
  CD16bright CD56dim, Month 24: number analyzed (Participants) | 170
  CD16bright CD56dim, Month 24 | -12.94 [-37.36 to 10.95]

ADVERSE EVENTS:
Time Frame: From baseline up to Month 45
Arm/Group | Experimental: Mavenclad®
All-Cause Mortality (participants affected / at risk) | 0/270
Serious Adverse Events (participants affected / at risk) | 14/270
Other Adverse Events (participants affected / at risk) | 225/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Mavenclad® (N=270)
Left ventricular dysfunction (Cardiac disorders) | 1
Diplopia (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Vestibular neuronitis (Infections and infestations) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Carotid endarterectomy (Surgical and medical procedures) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Ischaemic stroke (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Interspinous osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Mavenclad® (N=270)
Diarrhoea (Gastrointestinal disorders) | 26
Fatigue (General disorders) | 31
Nasopharyngitis (Infections and infestations) | 57
Urinary tract infection (Infections and infestations) | 32
Alopecia (Skin and subcutaneous tissue disorders) | 21
Nausea (Gastrointestinal disorders) | 31
Oral herpes (Infections and infestations) | 20
Upper respiratory tract infection (Infections and infestations) | 27
Lymphopenia (Blood and lymphatic system disorders) | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 30
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 17
Neck Pain (Musculoskeletal and connective tissue disorders) | 14
Pain in extrimity (Musculoskeletal and connective tissue disorders) | 22
Dizziness (Nervous system disorders) | 20
Headache (Nervous system disorders) | 87
Paraesthesia (Nervous system disorders) | 15
Anxiety (Psychiatric disorders) | 16
Insomnia (Psychiatric disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT03364036/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03364036/SAP_002.pdf